CLINICAL TRIAL: NCT00137423
Title: A Phase 2 Efficacy And Safety Study Of SU011248 Administered In A Continuous Daily Regimen In Patients With Cytokine-Refractory Metastatic Renal Cell Carcinoma
Brief Title: Study Of SU011248 (Sunitinib) Given In A Continuous Daily Regimen In Patients With Advanced Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181061
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Carcinoma, Renal Cell Metastasis
MeSH Terms: conditions — Carcinoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SU011248 (sunitinib) (Experimental): Single-arm study
  Interventions: Drug: SU011248 (sunitinib)

INTERVENTIONS:
Drug: SU011248 (sunitinib) — 37.5 mg/day, oral, continuous daily dosing

SUMMARY:
To evaluate the anti-tumor activity of SU011248 (sunitinib) in cytokine-refractory metastatic renal cell carcinoma (RCC) when administered in a continuous treatment regimen

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven renal cell carcinoma with metastases.
* Evidence of unidimensionally measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST).
* Failure of 1 prior cytokine-based therapy for metastatic disease. Patients treated with IFN-á alone must have received IFN-á for at least 4 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Resolution of all acute toxic effects of prior therapy or surgical procedures to grade 1.
* Adequate organ function

Exclusion Criteria:

* Prior treatment with any systemic therapy other than 1 cytokine-based therapy.
* Previous treatment on a SU011248 (sunitinib) clinical trial.
* Major surgery, radiation therapy, or systemic therapy within 4 weeks of starting the study treatment.
* Diagnosis of any second malignancy within the last 3 years, except basal cell carcinoma, squamous cell skin cancer, or in situ carcinoma that has been adequately treated with no evidence of recurrent disease for 12 months.
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease on screening Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) scan.
* Any of the following within the 12 months prior to starting the study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of grade 2, atrial fibrillation of any grade, or QTc interval >450 msec for males or >470 msec for females.
* Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy).
* Ongoing treatment with therapeutic doses of Coumadin (however, low dose Coumadin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
* Known human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2005-05; Primary Completion 2007-09 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (2):
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Las Vegas, Nevada
- Pfizer Investigational Site, Villejuif, France
- Germany (2):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, München
- Pfizer Investigational Site, Thessaloniki, Greece
- Pfizer Investigational Site, Nijmegen, Gelderland, Netherlands
- Sweden (2):
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Stockholm
- Pfizer Investigational Site, Sankt Gallen, Switzerland

REFERENCES:
- [Derived] de Velasco G, McKay RR, Lin X, Moreira RB, Simantov R, Choueiri TK. Comprehensive Analysis of Survival Outcomes in Non-Clear Cell Renal Cell Carcinoma Patients Treated in Clinical Trials. Clin Genitourin Cancer. 2017 Dec;15(6):652-660.e1. doi: 10.1016/j.clgc.2017.03.004. Epub 2017 Mar 21. PMID 28410911
- [Derived] Grunwald V, Lin X, Kalanovic D, Simantov R. Early Tumour Shrinkage: A Tool for the Detection of Early Clinical Activity in Metastatic Renal Cell Carcinoma. Eur Urol. 2016 Dec;70(6):1006-1015. doi: 10.1016/j.eururo.2016.05.010. Epub 2016 May 26. PMID 27238653
- [Derived] Grunwald V, McKay RR, Krajewski KM, Kalanovic D, Lin X, Perkins JJ, Simantov R, Choueiri TK. Depth of remission is a prognostic factor for survival in patients with metastatic renal cell carcinoma. Eur Urol. 2015 May;67(5):952-8. doi: 10.1016/j.eururo.2014.12.036. Epub 2015 Jan 7. PMID 25577718
- [Derived] Escudier B, Roigas J, Gillessen S, Harmenberg U, Srinivas S, Mulder SF, Fountzilas G, Peschel C, Flodgren P, Maneval EC, Chen I, Vogelzang NJ. Phase II study of sunitinib administered in a continuous once-daily dosing regimen in patients with cytokine-refractory metastatic renal cell carcinoma. J Clin Oncol. 2009 Sep 1;27(25):4068-75. doi: 10.1200/JCO.2008.20.5476. Epub 2009 Aug 3. PMID 19652072
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181061&StudyName=Study%20Of%20SU011248%20Given%20In%20A%20Continuous%20Daily%20Regimen%20In%20Patients%20With%20Advanced%20Renal%20Cell%20Cancer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients must have failed 1 prior cytokine-based therapy for metastatic renal cell carcinoma and had to have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
Pre-assignment Details: ECOG performance status definition 0=fully active, able to carry on all pre-disease activities without restriction 1= restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature (eg light house work or office work)
Groups:
- AM Dose Sunitinib Malate (SU011248): Patients received a starting dose of 37.5 mg/day of sunitinib malate in the morning repeated 4-week cycles continuing for up to 1 year in absence of any withdrawal criteria.Per the statistical analysis plan, the primary outcome of objective response was evaluated in patients who had measurable disease at baseline, the correct histological cancer type, & were refractory to prior cytokine-based therapy. Of 107 subjects enrolled, 2 patients did not have measurable disease at baseline, and therefore, were excluded from the analysis.
- PM Dose Sunitinib Malate (SU011248): Patients received a starting dose of 37.5 mg/day of sunitinib malate in the evening repeated 4-week cycles continuing for up to 1 year in absence of any withdrawal criteria.Per the statistical analysis plan, the primary outcome of objective response was evaluated in patients who had measurable disease at baseline, the correct histological cancer type, & were refractory to prior cytokine-based therapy. Of 107 subjects enrolled, 2 patients did not have measurable disease at baseline, and therefore, were excluded from the analysis.
Period: Overall Study
Arm/Group | AM Dose Sunitinib Malate (SU011248) | PM Dose Sunitinib Malate (SU011248)
Started | 54 | 53
Completed | 15 | 9
Not Completed | 39 | 44
Not completed — Adverse Event | 7 | 9
Not completed — consent withdrawn | 1 | 1
Not completed — Lack of Efficacy | 31 | 33
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AM Dose Sunitinib Malate (SU011248) | PM Dose Sunitinib Malate (SU011248) | Total
Number analyzed (Participants) | 54 | 53 | 107
Age Continuous [Mean (Standard Deviation); unit: years] | 59.3 (9.27) | 57.2 (11.48) | 58.2 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 46 | 42 | 88

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Complete Response[CR] + Partial Response[PR]) in Subjects
Description: Confirmed objective responses using RECIST criteria defined as responses persisting on repeat imaging study for 2 assessments with at least 4 weeks between, and evaluating all target and non-target sites followed since baseline. Two PRs separated by an SD or NE visit in between was considered a confirmed response if the 2 PRs were > 4 weeks apart. CR=disappearance of all target lesions. PR is a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: 4 week treatment cycles up to 1 year in absence of withdrawal criteria requiring discontinuation includes 28 day post study follow up
Population: ITT; CR,PR calculated from patients with measurable disease at baseline+correct histological cancer type+ refractory to prior cytokine-based therapy n= 53,52 (AM,PM)
Measure: Number; unit: participants
Groups:
- AM Dose Sunitinib Malate (SU011248): Patients received a starting dose of 37.5 mg/day of sunitinib malate in the morning repeated 4-week cycles continuing for up to 1 year in absence of any withdrawal criteria.
- PM Dose Sunitinib Malate (SU011248): Patients received a starting dose of 37.5 mg/day of sunitinib malate in the evening repeated 4-week cycles continuing for up to 1 year in absence of any withdrawal criteria.
Arm/Group | AM Dose Sunitinib Malate (SU011248) | PM Dose Sunitinib Malate (SU011248)
Number analyzed (Participants) | 54 | 53
participants | 15 | 6
Statistical Analysis 1: Comparison: AM Dose Sunitinib Malate (SU011248); Objective response rate required a sample size of 100 to test null hypothesis that true response rate was <=5% versus alternative hypothesis that true response rate was >=15% with 90% power and alpha level of 0.05. If number of OR> =11 null hypothesis that true response rate was <=5% could be rejected with a target α error rate of 0.05; Test type: Superiority or Other; F distribution; Objective Response Rate = 28.3, 95% CI [16.8 to 42.3]
Statistical Analysis 2: Comparison: PM Dose Sunitinib Malate (SU011248); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; F distribution; Objective Response Rate = 11.5, 95% CI [4.4 to 23.4]

2. Secondary Outcome: Duration of Tumor Response
Description: Using RECIST criteria: date of 1st objective tumor response (CR or PR) subsequently confirmed to date of 1st objective tumor progression or to death due to any cause within 28 days after last dose of study medication, whichever was first. Censored on day after the date of the last oncologic assessment documenting no tumor progression.
Time Frame: as for outcome 1
Population: ITT; DR time from start of 1st documentation of objective tumor response to 1st documentation of objective tumor progression or death & calculated for the subgroup of subjects with a confirmed objective tumor response. Descriptive statistics for responders who had an event. Total number responders n= 15,6(AM,PM). Response duration n=7,3(AM,PM).
Measure: Median (Full Range); unit: weeks
Arm/Group | AM Dose Sunitinib Malate (SU011248) | PM Dose Sunitinib Malate (SU011248)
Number analyzed (Participants) | 54 | 53
weeks | 24.0 [16.1 to 64.1] | 32.0 [16.1 to 32.1]

3. Secondary Outcome: Time to Tumor Progression (TTP)
Description: Time from date of first dose of study medication to date of first documentation of objective tumor progression using RECIST criteria that occurred on treatment including within 28 days after the last dose of study medication. TTP censored on the day following the date of last oncologic assessment documenting absence of tumor progression. TTP based on the number of subjects with measurable disease at baseline, the correct histological cancer type, and had disease that was refractory to prior cytokine-based therapy(105 in total group).
Time Frame: as for outcome 1
Population: ITT;TTP calculated based on subgroup with baseline disease assessment, measurable disease at baseline, correct histological type and refractory to cytokine.Estimates based on Kaplan-Meier method with 95% CI calculated based on Brookmeyer and Crowley. n=53,52(AM,PM).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | AM Dose Sunitinib Malate (SU011248) | PM Dose Sunitinib Malate (SU011248)
Number analyzed (Participants) | 54 | 53
weeks | 35.7 [27.9 to 50.0] | 35.9 [20.3 to 38.1]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Using RECIST criteria: Time from date 1st dose study medication to date 1st documentation of objective tumor progression or death due to any cause occurring on treatment including within 28 days after last dose, whichever occurred 1st. Censored on day following the date of last oncologic assessment documenting absence of tumor progression. PFS based on the number of subjects with measurable disease at baseline, the correct histological cancer type, and had disease that was refractory to prior cytokine-based therapy(105 in total group).
Time Frame: as for outcome 1
Population: ITT; Calculation based on subgroup of patients with baseline disease assessment, measurable disease at baseline, correct histological type and are refractory to cytokine. Estimates based on Kaplan-Meier method with 95% CI calculated based on Brookmeyer and Crowley. N=53,52(AM,PM).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | AM Dose Sunitinib Malate (SU011248) | PM Dose Sunitinib Malate (SU011248)
Number analyzed (Participants) | 54 | 53
weeks | 35.7 [27.6 to 50.0] | 35.3 [20.3 to 38.1]

5. Secondary Outcome: Overall Survival
Description: Overall survival is time from the date of first dose of medication to the date of death due to any cause
Time Frame: as for outcome 1
Population: ITT; Patients who are alive at the time of analysis or who are lost to follow up are censored on the last date they were known to be alive. Estimates are based on the Kaplan-Meier method with 95% CI calculated based on Brookmeyer and Crowley method. n=54,53(AM,PM).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | AM Dose Sunitinib Malate (SU011248) | PM Dose Sunitinib Malate (SU011248)
Number analyzed (Participants) | 54 | 53
weeks | 91.4 [69.4 to 115.4] | 76.4 [59.6 to 108.3]
Statistical Analysis 1: Comparison: AM Dose Sunitinib Malate (SU011248); Test type: Superiority or Other; Kaplan-Meier method; 1-year survival rate = 77.4, 95% CI [63.6 to 86.5] — valid presentation only if at least 1 patient has overall survival >=1 year. Based on normal approximation, 95% CI will be derived by log transformation of the cumulative hazard rate
Statistical Analysis 2: Comparison: PM Dose Sunitinib Malate (SU011248); Test type: Superiority or Other; Kaplan-Meier method; 1-year survival rate = 66.0, 95% CI [51.6 to 77.1] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Summary of FACIT Fatigue Scale Overall Score
Description: FACIT Fatigue Scale: Overall score from 13-questionnaire, which measures fatigue / asthenia for patients with chronic, life-threatening illnesses. For each question, a patient rates his / her condition for the past week on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). Higher scores always represent less fatigue / asthenia. Outcome based on completed questionnaires.
Time Frame: Day 1 and day 15 of each treatment cycle from cycle 1 to cycle 4; day 1 of each treatment cycle after cycle 4 up to one year.
Population: ITT; Results summarized by cohort & time point through Cycle 13 (the last cycle for which more than 3 subjects completed the questionnaire on either arm). If more than 50% of the items in the scale were answered, then missing items were imputed with the mean of the non-missing items scored at that visit. Outcome based on completed questionnaires.
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- AM Dose Sunitinib Malate: Patients received a starting dose of 37.5 mg/day of sunitinib malate in the morning repeated 4-week cycles continuing for up to 1 year in absence of any withdrawal criteria.
- PM Dose Sunitinib Malate: Patients received a starting dose of 37.5 mg/day of sunitinib malate in the evening repeated 4-week cycles continuing for up to 1 year in absence of any withdrawal criteria.Per the statistical analysis plan, the primary outcome of objective response was evaluated in patients who had measurable disease at baseline, the correct histological cancer type, & were refractory to prior cytokine-based therapy. Of 107 subjects enrolled, 2 patients did not have measurable disease at baseline, and therefore, were excluded from the analysis.
Arm/Group | AM Dose Sunitinib Malate | PM Dose Sunitinib Malate
Number analyzed (Participants) | 54 | 53
score on scale
  Baseline Score n=52,52 | 39.5 (11.41) | 39.6 (10.15)
  Maximum Post-Baseline Score n=53,52 | 43.4 (7.86) | 42.7 (8.19)
  Minimum Post-Baseline Score n=53,52 | 28.0 (12.34) | 29.4 (13.65)

7. Secondary Outcome: Change From Baseline in Euro-QoL Five Dimension (EQ-5D) Weighted Health Index
Description: EQ-5D health status in 5 dimensions (mobility, self-care, pain / discomfort, anxiety / depression, usual activities) with a weighted health index based on general population values where 0.0=death and 1.0 = perfect health. Change: median index score at observation minus median index score at baseline.
Time Frame: as for outcome 6
Population: ITT
Measure: Median (Full Range); unit: score on scale
Arm/Group | AM Dose Sunitinib Malate (SU011248) | PM Dose Sunitinib Malate (SU011248)
Number analyzed (Participants) | 54 | 53
score on scale
  Maximum Increase | 0.0 [-0.7 to 0.9] | 0.0 [-0.3 to 1.0]
  Maximum Decrease | 0.0 [-0.8 to 0.8] | -0.1 [-0.6 to 0.7]

8. Secondary Outcome: Change From Baseline in EuroQoL Visual Analog Scale (EQ-VAS) Overall Health Thermometer Score
Description: EQ-VAS score on the self-rated "thermometer" indicated the patient's own assessment of their health status from 0 (worst) to 100 (best) imaginable health state. Change: median score at observation minus median score at baseline. Maximum changes (increase or decrease from baseline).
Time Frame: as for outcome 6
Population: ITT
Measure: Median (Full Range); unit: score on scale
Arm/Group | AM Dose Sunitinib Malate (SU011248) | PM Dose Sunitinib Malate (SU011248)
Number analyzed (Participants) | 54 | 53
score on scale
  Maximum Increase | 0.0 [-40.0 to 32.0] | 0.0 [-45.0 to 92.0]
  Maximum Decrease | -10.0 [-51.0 to 80.0] | -9.0 [-40.0 to 44.0]

ADVERSE EVENTS:
Arm/Group | AM Dose Sunitinib Malate (SU011248) | PM Dose Sunitinib Malate (SU011248)
Serious Adverse Events (participants affected / at risk) | 21 | 20
Other Adverse Events (participants affected / at risk) | 54 | 53
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | AM Dose Sunitinib Malate (SU011248) | PM Dose Sunitinib Malate (SU011248)
Thrombocytopenia (Blood and lymphatic system disorders) | 3/54 | 1/53
Anaemia (Blood and lymphatic system disorders) | 1/54 | 2/53
Cardiac arrest (Cardiac disorders) | 0/54 | 1/53
Cardiac failure congestive (Cardiac disorders) | 0/54 | 1/53
Vertigo (Ear and labyrinth disorders) | 1/54 | 0/53
Eye pain (Eye disorders) | 0/54 | 1/53
Abdominal pain (Gastrointestinal disorders) | 4/54 | 3/53
Haematemesis (Gastrointestinal disorders) | 1/54 | 2/53
Vomiting (Gastrointestinal disorders) | 2/54 | 1/53
Nausea (Gastrointestinal disorders) | 0/54 | 2/53
Oesophagitis (Gastrointestinal disorders) | 1/54 | 1/53
Subileus (Gastrointestinal disorders) | 2/54 | 0/53
Constipation (Gastrointestinal disorders) | 0/54 | 1/53
Diarrhoea (Gastrointestinal disorders) | 0/54 | 1/53
Gastritis haemorrhagic (Gastrointestinal disorders) | 0/54 | 1/53
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/54 | 0/53
Melaena (Gastrointestinal disorders) | 1/54 | 0/53
Pancreatitis acute (Gastrointestinal disorders) | 1/54 | 0/53
Salivary hypersecretion (Gastrointestinal disorders) | 1/54 | 0/53
Stomatitis (Gastrointestinal disorders) | 1/54 | 0/53
Asthenia (General disorders) | 1/54 | 2/53
Disease progression (General disorders) | 0/54 | 3/53
Fatigue (General disorders) | 0/54 | 2/53
Gait disturbance (General disorders) | 1/54 | 1/53
Mucosal inflammation (General disorders) | 2/54 | 0/53
Oedema peripheral (General disorders) | 2/54 | 0/53
Pyrexia (General disorders) | 0/54 | 2/53
Hypothermia (General disorders) | 1/54 | 0/53
Multi-organ failure (General disorders) | 1/54 | 0/53
Organ failure (General disorders) | 0/54 | 1/53
Performance status decreased (General disorders) | 0/54 | 1/53
Cholangitis acute (Hepatobiliary disorders) | 1/54 | 0/53
Perirectal abscess (Infections and infestations) | 1/54 | 1/53
Pneumonia (Infections and infestations) | 1/54 | 0/53
Respiratory tract infection (Infections and infestations) | 1/54 | 0/53
Sepsis (Infections and infestations) | 1/54 | 0/53
Urinary tract infection (Infections and infestations) | 1/54 | 0/53
Burn oesophageal (Injury, poisoning and procedural complications) | 1/54 | 0/53
Fall (Injury, poisoning and procedural complications) | 1/54 | 0/53
Wound (Injury, poisoning and procedural complications) | 1/54 | 0/53
Aspiration pleural cavity (Investigations) | 1/54 | 0/53
Blood creatinine increased (Investigations) | 0/54 | 1/53
Anorexia (Metabolism and nutrition disorders) | 1/54 | 3/53
Dehydration (Metabolism and nutrition disorders) | 1/54 | 3/53
Hyperkalaemia (Metabolism and nutrition disorders) | 1/54 | 1/53
Hypoglycaemia (Metabolism and nutrition disorders) | 1/54 | 1/53
Diabetes mellitus (Metabolism and nutrition disorders) | 1/54 | 0/53
Hypercalcaemia (Metabolism and nutrition disorders) | 0/54 | 1/53
Hyperglycaemia (Metabolism and nutrition disorders) | 1/54 | 0/53
Hypernatraemia (Metabolism and nutrition disorders) | 0/54 | 1/53
Hyponatraemia (Metabolism and nutrition disorders) | 0/54 | 1/53
Malnutrition (Metabolism and nutrition disorders) | 1/54 | 0/53
Bone lesion (Musculoskeletal and connective tissue disorders) | 1/54 | 0/53
Flank pain (Musculoskeletal and connective tissue disorders) | 0/54 | 1/53
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1/54 | 0/53
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1/54 | 0/53
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/54 | 0/53
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/54 | 0/53
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/54 | 1/53
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/54 | 1/53
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/54 | 1/53
Dizziness (Nervous system disorders) | 2/54 | 1/53
Syncope (Nervous system disorders) | 0/54 | 2/53
Brain oedema (Nervous system disorders) | 0/54 | 1/53
Cerebrovascular accident (Nervous system disorders) | 0/54 | 1/53
Depressed level of consciousness (Nervous system disorders) | 1/54 | 0/53
Dysaesthesia (Nervous system disorders) | 1/54 | 0/53
Paresis (Nervous system disorders) | 1/54 | 0/53
Peripheral sensory neuropathy (Nervous system disorders) | 0/54 | 1/53
Confusional state (Psychiatric disorders) | 1/54 | 1/53
Anuria (Renal and urinary disorders) | 2/54 | 0/53
Urinary retention (Renal and urinary disorders) | 1/54 | 1/53
Haematuria (Renal and urinary disorders) | 0/54 | 1/53
Obstructive uropathy (Renal and urinary disorders) | 1/54 | 0/53
Renal failure (Renal and urinary disorders) | 0/54 | 1/53
Renal failure acute (Renal and urinary disorders) | 0/54 | 1/53
Renal haemorrhage (Renal and urinary disorders) | 0/54 | 1/53
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/54 | 0/53
Pelvic pain (Reproductive system and breast disorders) | 1/54 | 0/53
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/54 | 1/53
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2/54 | 0/53
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2/54 | 0/53
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/54 | 0/53
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0/54 | 1/53
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0/54 | 1/53
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1/54 | 0/53
Pleurodesis (Surgical and medical procedures) | 1/54 | 0/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | AM Dose Sunitinib Malate (SU011248) | PM Dose Sunitinib Malate (SU011248)
Anaemia (Blood and lymphatic system disorders) | 7/54 | 9/53
Thrombocytopenia (Blood and lymphatic system disorders) | 8/54 | 6/53
Neutropenia (Blood and lymphatic system disorders) | 5/54 | 7/53
Leukopenia (Blood and lymphatic system disorders) | 3/54 | 3/53
Vertigo (Ear and labyrinth disorders) | 4/54 | 3/53
Diarrhoea (Gastrointestinal disorders) | 41/54 | 40/53
Stomatitis (Gastrointestinal disorders) | 25/54 | 21/53
Nausea (Gastrointestinal disorders) | 25/54 | 19/53
Dyspepsia (Gastrointestinal disorders) | 22/54 | 15/53
Vomiting (Gastrointestinal disorders) | 16/54 | 18/53
Abdominal pain (Gastrointestinal disorders) | 14/54 | 13/53
Constipation (Gastrointestinal disorders) | 14/54 | 8/53
Abdominal pain upper (Gastrointestinal disorders) | 13/54 | 6/53
Oral pain (Gastrointestinal disorders) | 4/54 | 6/53
Flatulence (Gastrointestinal disorders) | 1/54 | 8/53
Glossodynia (Gastrointestinal disorders) | 5/54 | 3/53
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0/54 | 7/53
Haemorrhoids (Gastrointestinal disorders) | 4/54 | 3/53
Rectal haemorrhage (Gastrointestinal disorders) | 5/54 | 2/53
Dysphagia (Gastrointestinal disorders) | 2/54 | 4/53
Gingival bleeding (Gastrointestinal disorders) | 3/54 | 3/53
Asthenia (General disorders) | 24/54 | 20/53
Fatigue (General disorders) | 19/54 | 22/53
Mucosal inflammation (General disorders) | 16/54 | 9/53
Pyrexia (General disorders) | 9/54 | 10/53
Chest pain (General disorders) | 9/54 | 9/53
Oedema peripheral (General disorders) | 9/54 | 5/53
Chills (General disorders) | 4/54 | 3/53
Nasopharyngitis (Infections and infestations) | 6/54 | 4/53
Bronchitis (Infections and infestations) | 4/54 | 2/53
Oral herpes (Infections and infestations) | 3/54 | 3/53
Urinary tract infection (Infections and infestations) | 5/54 | 1/53
Weight decreased (Investigations) | 15/54 | 17/53
Blood lactate dehydrogenase increased (Investigations) | 6/54 | 2/53
Blood creatinine increased (Investigations) | 1/54 | 6/53
Blood alkaline phosphatase increased (Investigations) | 2/54 | 4/53
Anorexia (Metabolism and nutrition disorders) | 21/54 | 20/53
Dehydration (Metabolism and nutrition disorders) | 1/54 | 8/53
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 6/54 | 2/53
Hyperkalaemia (Metabolism and nutrition disorders) | 3/54 | 3/53
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11/54 | 11/53
Arthralgia (Musculoskeletal and connective tissue disorders) | 9/54 | 8/53
Back pain (Musculoskeletal and connective tissue disorders) | 8/54 | 6/53
Myalgia (Musculoskeletal and connective tissue disorders) | 2/54 | 8/53
Dysgeusia (Nervous system disorders) | 13/54 | 15/53
Headache (Nervous system disorders) | 6/54 | 8/53
Dizziness (Nervous system disorders) | 9/54 | 4/53
Ageusia (Nervous system disorders) | 4/54 | 7/53
Insomnia (Psychiatric disorders) | 4/54 | 8/53
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17/54 | 11/53
Cough (Respiratory, thoracic and mediastinal disorders) | 6/54 | 10/53
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8/54 | 6/53
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6/54 | 7/53
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 28/54 | 23/53
Hair colour changes (Skin and subcutaneous tissue disorders) | 18/54 | 20/53
Rash (Skin and subcutaneous tissue disorders) | 12/54 | 11/53
Dry skin (Skin and subcutaneous tissue disorders) | 10/54 | 12/53
Erythema (Skin and subcutaneous tissue disorders) | 11/54 | 8/53
Skin discolouration (Skin and subcutaneous tissue disorders) | 4/54 | 7/53
Alopecia (Skin and subcutaneous tissue disorders) | 6/54 | 3/53
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2/54 | 4/53
Pruritus (Skin and subcutaneous tissue disorders) | 1/54 | 5/53
Hypertension (Vascular disorders) | 25/54 | 23/53
Haemorrhage (Vascular disorders) | 4/54 | 4/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.